CLINICAL TRIAL: NCT01658176
Title: An Open-Label Randomized Phase 2 Study Of PF-04691502 (PI3K/mTOR Inhibitor) In Combination With Exemestane Compared With Exemestane Alone In Patients With Estrogen Receptor Positive, Her-2 Negative Advanced Breast Cancer
Brief Title: Study Of PF-04691502 (PI3K/mTOR Inhibitor) In Combination With Exemestane Compared With Exemestane Alone In Patients With Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1271005
Record Dates: First submitted 2012-07-16; First posted 2012-08-06 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Breast Neoplasms
Keywords: Estrogen receptor positive; Her-2 negative; advanced breast cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-amino-8-(4-(2-hydroxyethoxy)cyclohexyl)-6-(6-methoxypyridin-3-yl)-4-methylpyrido(2,3-d)pyrimidin-7(8H)-one; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04691502 + Exemestane (Experimental): PF-04691502 in combination with Exemestane
  Interventions: Drug: PF-04691502; Drug: Exemestane
- Exemestane (Active Comparator): Exemestane alone
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: PF-04691502 — PF-04691502 administered orally at 8 mg as a continuous daily dosing schedule
  Arms: PF-04691502 + Exemestane
Drug: Exemestane — Exemestane administered orally at 25 mg as a continuous daily dosing schedule
  Arms: PF-04691502 + Exemestane
Drug: Exemestane — Exemestane administered orally at 25 mg as a continuous daily dosing schedule
  Arms: Exemestane

SUMMARY:
PF-04691502 is an inhibitor of PI3K and mTOR kinase. Exemestane is an aromatase inhibitor for the treatment of advanced breast cancer in women whose disease has progressed following tamoxifen therapy. The combination of PF-04691502 and exemestane might mitigate resistance to hormonal therapy and result in greater clinical benefit than exemestane alone in women with estrogen receptor positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable estrogen receptor positive, Her-2 negative advanced breast cancer
* Previously treated with an aromatase inhibitor
* Primary or secondary hormone resistance
* Acceptable glucose control, bone marrow, liver and kidney function

Exclusion Criteria:

* Inflammatory breast carcinoma
* Prior therapy with an agent active on PI3K, Akt, and/or mTOR
* Known hypersensitivity to exemestane
* Significant gastrointestinal abnormalities which may impair intake, transit, or absorption of the study drugs
* Current or anticipated need for food or drugs that are known inhibitors or inducers of CYP3A4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Baseline up to month 12

SECONDARY OUTCOMES:
Objective tumor response using RECIST | Baseline up to month 12
Duration of tumor response | Baseline up to month 12
Clinical benefit response | Baseline up to month 12
Overall Survival | 2 years
Biomarkers related to PI3K/mTOR signal deregulation and markers of cellular proliferation and apoptosis in primary tumor tissue | Baseline
Maximum concentration (Cmax) of single dose of PF-04691502 | Day 2 Pre-dose, and 1 , 2, 4 and 24 hours post-dose
Maximum concentration (Cmax) of single dose exemestane | Day 1 pre-dose, and 1, 2, 4 and 24 hours post-dose
Maximum concentration (Cmax) of PF-04691502 and exemestane when administered in combination | Day 8 Pre-dose, and 1, 2, 4 and 24 hours post-dose, Weel 5, 9, 13, 17, 21, and 25
Pharmacodynamic endpoints including serum glucose, insulin, HbA1c, cholesterol and triglycerides | 12 months
Heath related quality of life measured by Functional Assessment of Cancer Therapy- Breast | 12 months
Area under the plasma concentration versus time curve (AUC) of single dose of PF-04691502 | Day 2 Pre-dose, and 1 , 2, 4 and 24 hours post-dose
Area under the plasma concentration versus time curve (AUC) of single dose exemestane | Day 1 pre-dose, and 1, 2, 4 and 24 hours post-dose
Area under the plasma concentration versus time curve (AUC) of PF-04691502 and exemestane when administered in combination | Day 8 Pre-dose, and 1, 2, 4 and 24 hours post-dose, Weel 5, 9, 13, 17, 21, and 25

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1271005&StudyName=Study%20Of%20PF-04691502%20%28PI3K/mTOR%20Inhibitor%29%20In%20Combination%20With%20Exemestane%20Compared%20With%20Exemestane%20Alone%20In%20Patients%20with%20Advanced%20Breas